CLINICAL TRIAL: NCT07161479
Title: A Multicenter, Randomized, Single-Blinded Trial Comparing Argon Plasma Coagulation and Endoscopic Mucosal Resection for Gastric Adenoma With Low-Grade Dysplasia
Brief Title: Argon Plasma Coagulation Versus Endoscopic Mucosal Resection for Gastric Adenoma (CLER-GA)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Collaborators: Samsung Medical Center, Sungkyunkwan University School of Medicine (Unknown)
Responsible Party: Principal Investigator, Hyuk Lee, Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SMC 2025-04-026-001
Record Dates: First submitted 2025-08-30; First posted 2025-09-08 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-08

CONDITIONS: Gastric Adenoma; Stomach Neoplasms; Precancerous Conditions; Dysplasia Stomach
Keywords: Gastric adenoma; Low-grade dysplasia; Precancerous gastric lesion; Argon plasma coagulation (APC); Endoscopic mucosal resection (EMR); Endoscopic therapy; Local recurrence; Randomized controlled trial; Stomach neoplasms
MeSH Terms: conditions — Stomach Neoplasms; Precancerous Conditions | interventions — Argon Plasma Coagulation; Endoscopic Mucosal Resection

STUDY DESIGN:
Intervention Model Description: This is a multicenter, randomized, single-blinded, parallel assignment trial. Eligible participants with gastric adenomas ≤ 1 cm will be randomly assigned in a 1:1 ratio to undergo either argon plasma coagulation (APC) or endoscopic mucosal resection (EMR). Patients will be blinded to treatment allocation, while treating endoscopists cannot be blinded due to the nature of the procedures.
Who Masked: Participant
Masking Description: Participants are blinded to the treatment allocation. Due to the nature of the procedures, endoscopists performing APC or EMR cannot be blinded. Outcome assessments are based on objective endoscopic and histologic findings, and therefore independent masking of assessors was not applied.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Argon Plasma Coagulation (APC) (Experimental): Participants undergo argon plasma coagulation for gastric adenoma ≤ 1 cm.
  Interventions: Procedure: Argon Plasma Coagulation (APC)
- Endoscopic Mucosal Resection (EMR) (Active Comparator): Participants undergo endoscopic mucosal resection for gastric adenoma ≤ 1 cm.
  Interventions: Procedure: Endoscopic Mucosal Resection (EMR)

INTERVENTIONS:
Procedure: Argon Plasma Coagulation (APC) — Ablation of gastric adenoma using argon plasma coagulation.
  Arms: Argon Plasma Coagulation (APC)
Procedure: Endoscopic Mucosal Resection (EMR) — Endoscopic resection of gastric adenoma by mucosal resection technique.
  Arms: Endoscopic Mucosal Resection (EMR)

SUMMARY:
Gastric adenomas with low-grade dysplasia (LGD) are considered precancerous lesions of the stomach. While these lesions carry a lower risk of progressing to gastric cancer compared with high-grade dysplasia, there is still uncertainty about the best way to manage them. International medical guidelines differ in their recommendations, and for very small lesions (1 cm or smaller), some guidelines provide no clear direction. This creates uncertainty for both patients and physicians about whether to treat these lesions or simply observe them over time.

Two endoscopic treatment methods are widely used in clinical practice: endoscopic mucosal resection (EMR) and argon plasma coagulation (APC). EMR involves lifting and cutting out the lesion. Its major advantage is that it removes the lesion completely and allows for detailed pathological examination. However, EMR can be technically more demanding, takes more time, and may carry higher risks of complications such as bleeding or perforation. It also usually involves higher medical costs.

In contrast, APC is a technique that uses ionized argon gas and electrical current to coagulate tissue without direct contact. APC is simpler to perform, takes less time, and is generally less invasive. Patients undergoing APC may have shorter hospital stays, lower costs, and fewer complications. However, APC does not provide a specimen for pathology, so complete removal of the lesion cannot be confirmed. This means there is a possibility of local recurrence.

Several retrospective studies have examined APC for gastric LGD, and results have suggested it may be effective for small lesions. However, recurrence rates reported in previous studies have varied widely, from less than 2% to more than 20%. Importantly, no large randomized controlled trial has directly compared APC with EMR for small gastric LGD lesions. This study seeks to fill that gap.

The goal of this clinical trial is to compare the effectiveness and safety of APC and EMR for treating gastric adenomas that are 1 cm or smaller with low-grade dysplasia. Specifically, the study aims to determine whether APC is "non-inferior" to EMR in preventing local recurrence of these lesions. In other words, researchers want to know if APC works just as well as EMR in controlling the disease, while also offering potential advantages such as fewer complications, shorter procedure time, and lower costs.

Participants in this study will:

Be adults (age 20 or older) diagnosed with a gastric adenoma 1 cm or smaller with low-grade dysplasia.

Be randomly assigned (by chance, like flipping a coin) to receive either APC or EMR.

Receive standard medical care after the procedure, including medications to help the stomach heal.

Return for follow-up endoscopy at 3 months and 12 months after the procedure. During these visits, the treated area will be checked carefully, and biopsies may be taken to determine whether the lesion has recurred.

Provide information about any complications, the duration of the procedure, and their recovery experience.

The main question is whether APC can prevent recurrence of gastric adenomas as effectively as EMR. Secondary questions include how the two treatments differ in terms of complications (such as bleeding or perforation) and procedure time.

Both APC and EMR are already established and commonly used treatments for gastric lesions. By directly comparing these two methods in a randomized controlled trial, this study will provide important evidence to guide future recommendations for patients with small gastric adenomas. The findings may help physicians and patients choose the best treatment option, balancing safety, effectiveness, and convenience.

DETAILED DESCRIPTION:
Gastric adenomas with low-grade dysplasia (LGD) represent precancerous changes in the stomach lining. Unlike high-grade dysplasia (HGD), which carries a well-established high risk of progression to gastric cancer and is uniformly recommended for endoscopic resection, LGD has a much lower risk of malignant transformation. Some long-term follow-up studies suggest that fewer than 10% of LGD lesions progress to cancer within five years. As a result, there has been longstanding debate over whether LGD lesions, particularly those measuring 1 cm or smaller, should be actively treated or only monitored.

International guidelines differ on this issue. The Vienna classification recommends either endoscopic resection or close surveillance. The American Society of Gastrointestinal Endoscopy (ASGE) guidelines do not provide explicit recommendations for LGD, focusing instead on HGD and cancer. The British Society of Gastroenterology (BSG) advises complete removal of adenomas but without specifying the method. Only the updated European Society of Gastrointestinal Endoscopy (ESGE) guideline explicitly recommends endoscopic mucosal resection (EMR) for lesions smaller than 1 cm, while larger or suspicious lesions should be treated with endoscopic submucosal dissection (ESD). In contrast, Japanese and Korean gastric cancer guidelines primarily address early gastric cancer and provide no guidance specific to adenomas.

Currently, EMR and ESD are considered standard resection techniques. EMR is suitable for small, superficial lesions and allows en bloc removal with pathological confirmation, but it involves technical demands, longer procedure time, higher risk of complications, and greater costs. ESD extends these advantages to larger or fibrotic lesions but is even more technically demanding. In comparison, argon plasma coagulation (APC) is a non-contact ablative method using ionized argon gas to deliver high-frequency current. APC has been widely applied in therapeutic endoscopy for hemostasis and tissue ablation. It is technically simple, quicker, less invasive, and associated with fewer complications and lower costs. However, APC does not yield a resection specimen, making it impossible to confirm complete removal histologically, and the possibility of local recurrence remains.

Several retrospective studies have evaluated APC for gastric LGD, reporting local recurrence rates ranging from 1.7% to over 20%. The largest cohort suggested a recurrence rate of 2.6% for lesions ≤1 cm, compared to higher recurrence for 1-2 cm lesions. These results suggest that APC may be suitable for selected small LGD lesions, but the lack of randomized controlled trials (RCTs) leaves considerable uncertainty. Importantly, no RCT has directly compared APC with EMR, the standard resection method, in this specific population.

This study is therefore designed as a multicenter, randomized, single-blinded, controlled trial to evaluate whether APC is non-inferior to EMR in preventing local recurrence of gastric adenomas with LGD measuring 1 cm or smaller. A total of 160 adult participants will be enrolled across multiple academic hospitals in Korea. Eligible patients will be randomized 1:1 to receive either APC or EMR. Standard post-procedure management will be provided to all patients, including fasting, acid suppression, and routine monitoring. Participants will be followed for at least 12 months, with surveillance endoscopies scheduled at 3 months and 12 months to assess the treated site and obtain biopsies when indicated.

The primary endpoint is local recurrence rate at 12 months, defined as histological confirmation of LGD at the treated site. Secondary endpoints include overall procedure outcomes (complete ablation or en bloc resection), procedure-related complications (bleeding, perforation), procedure time, and hospitalization outcomes. Statistical analysis will follow both intention-to-treat and per-protocol principles, with non-inferiority margins prespecified.

Both APC and EMR are already established in routine practice and are not investigational devices in the United States. This trial does not involve an FDA IND or IDE. The significance of this study lies in generating high-quality prospective evidence that can directly inform clinical decision-making for patients with gastric LGD. If APC proves to be non-inferior to EMR, it could provide a simpler, less invasive, and more cost-effective alternative for selected patients with small adenomas, reducing procedure time and complication risk while maintaining effectiveness in preventing recurrence. Conversely, if APC shows inferior outcomes, it would reinforce EMR as the standard of care.

This study addresses an important knowledge gap in the management of gastric LGD and has potential to influence future guideline recommendations worldwide.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 20 years or older
* Diagnosed with gastric adenoma with low-grade dysplasia measuring ≤ 1 cm on endoscopy
* Scheduled to undergo endoscopic treatment
* Able and willing to provide written informed consent

Exclusion Criteria:

* Previous treatment for gastric adenoma or gastric cancer
* History of gastrectomy
* Diagnosis of gastric cancer or high-grade dysplasia at the time of enrollment
* Presence of multiple gastric adenomas
* Pregnant, breastfeeding, or possibility of pregnancy
* Uncontrolled chronic illnesses that may interfere with trial participation (e.g., uncontrolled hypertension, uncontrolled diabetes, chronic kidney disease, ascites, heart failure, psychiatric disorders)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2026-01-20 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Local recurrence rate of gastric adenoma with low-grade dysplasia | 12 months after treatment
  Proportion of participants with histologically confirmed recurrence of gastric adenoma at the treated site, as determined by follow-up endoscopy and biopsy.

SECONDARY OUTCOMES:
Procedure outcomes | At the time of index procedure
  Proportion of participants with complete ablation by APC or en bloc resection by EMR.
Procedure-related bleeding | Within 4 weeks after treatment
  Proportion of participants with bleeding defined as a hemoglobin decrease >2 g/dL accompanied by hematemesis, melena, or hypotension, occurring within 4 weeks of treatment.
Procedure-related perforation | Within 4 weeks after treatment
  Proportion of participants with perforation, defined as direct endoscopic evidence during the procedure or free air detected on chest radiograph after the procedure. Subcategories include gross perforation and microscopic perforation.
Procedure time | At the time of index procedure
  Average duration of the endoscopic procedure (APC or EMR), measured in minutes and seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Hyuk Lee, MD, PhD, Principal Investigator — Samsung Medical Center; Hyo-Joon Yang, MD, PhD, Principal Investigator — Kangbuk Samsung Hospital; Young-Il Kim, MD, PhD, Principal Investigator — National Cancer Center; Jong Yeul Lee, MD, PhD, Principal Investigator — National Cancer Center
Locations (3):
- South Korea (3):
  - National Cancer Center, Goyang-si
  - Kangbuk Samsung hospital, Seoul
  - Samsung Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: Yes
De-identified data may be shared upon reasonable request
Supporting Information: Study Protocol, SAP
Time Frame: De-identified individual participant data (IPD) and supporting documents will be made available beginning 6 months after publication of the main study results and will be accessible for up to 3 years thereafter.
Access Criteria: De-identified individual participant data (IPD) and supporting information (study protocol, statistical analysis plan) will be made available to qualified researchers affiliated with academic or medical institutions. Interested researchers must submit a written proposal describing the intended use of the data. Access will be granted after review and approval by the principal investigator. A data use agreement must be signed prior to release. Data will be shared through a secure institutional platform or by direct request to the principal investigator.

REFERENCES:
- [Result] Kim IH, Kang SJ, Choi W, Seo AN, Eom BW, Kang B, Kim BJ, Min BH, Tae CH, Choi CI, Lee CK, An HJ, Byun HK, Im HS, Kim HD, Cho JH, Pak K, Kim JJ, Bae JS, Yu JI, Lee JW, Choi J, Kim JH, Choi M, Jung MR, Seo N, Eom SS, Ahn S, Kim SJ, Lee SH, Lim SH, Kim TH, Han HS; Development Working Group for the Korean Practice Guideline for Gastric Cancer 2024 Task Force Team. Korean Practice Guidelines for Gastric Cancer 2024: An Evidence-based, Multidisciplinary Approach (Update of 2022 Guideline). J Gastric Cancer. 2025 Jan;25(1):5-114. doi: 10.5230/jgc.2025.25.e11. PMID 39822170
- [Result] Pimentel-Nunes P, Libanio D, Bastiaansen BAJ, Bhandari P, Bisschops R, Bourke MJ, Esposito G, Lemmers A, Maselli R, Messmann H, Pech O, Pioche M, Vieth M, Weusten BLAM, van Hooft JE, Deprez PH, Dinis-Ribeiro M. Endoscopic submucosal dissection for superficial gastrointestinal lesions: European Society of Gastrointestinal Endoscopy (ESGE) Guideline - Update 2022. Endoscopy. 2022 Jun;54(6):591-622. doi: 10.1055/a-1811-7025. Epub 2022 May 6. PMID 35523224
- [Result] Zhao G, Xue M, Hu Y, Lai S, Chen S, Wang L. How Commonly Is the Diagnosis of Gastric Low Grade Dysplasia Upgraded following Endoscopic Resection? A Meta-Analysis. PLoS One. 2015 Jul 16;10(7):e0132699. doi: 10.1371/journal.pone.0132699. eCollection 2015. PMID 26182344
- [Result] Cho SJ, Choi IJ, Kim CG, Lee JY, Kook MC, Park S, Ryu KW, Lee JH, Kim YW. Risk of high-grade dysplasia or carcinoma in gastric biopsy-proven low-grade dysplasia: an analysis using the Vienna classification. Endoscopy. 2011 Jun;43(6):465-71. doi: 10.1055/s-0030-1256236. Epub 2011 Mar 21. PMID 21425043
- [Result] Jung SJ, Cho SJ, Choi IJ, Kook MC, Kim CG, Lee JY, Park SR, Lee JH, Ryu KW, Kim YW. Argon plasma coagulation is safe and effective for treating smaller gastric lesions with low-grade dysplasia: a comparison with endoscopic submucosal dissection. Surg Endosc. 2013 Apr;27(4):1211-8. doi: 10.1007/s00464-012-2577-9. Epub 2012 Oct 18. PMID 23076459